CLINICAL TRIAL: NCT04396509
Title: Effects of Type of Delivery Mode and Gestational Age on Maternal Bonding
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: mai-nsd-c/s
Record Dates: First submitted 2020-05-16; First posted 2020-05-20 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Mother-Infant Interaction; Postnatal Depression; Postpartum Anxiety
Keywords: The Maternal Attachment Inventory; Postnatal Depression; Postpartum Anxiety
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women giving birth by normal vaginal delivery: 100 women delivered vaginally. . They were examined three month after delivery using Maternal Attachment Inventory (MAI) and a detailed history was taken. Women aged 18 to 45 years who delivered at term and had natural pregnancy (without any ART method),
  Interventions: Behavioral: Maternal Attachment Inventory Score
- women giving birth by c-section: 100 delivered with cesarean section. They were examined three month after delivery using Maternal Attachment Inventory (MAI) and a detailed history was taken. Women aged 18 to 45 years who delivered at term and had natural pregnancy (without any ART method),
  Interventions: Behavioral: Maternal Attachment Inventory Score

INTERVENTIONS:
Behavioral: Maternal Attachment Inventory Score — three month after delivery using Maternal Attachment Inventory (MAI) and a detailed history was taken.

SUMMARY:
To evaluate the effects of gestational age and other factors on maternal attachment relationship. There are different results in studies examining the effects of birth type on postpartum depression and mother-infant interaction. The aim of this study was to evaluate factors which affected mother-infant bond (MIB) using maternal attachment inventory (MAI).

DETAILED DESCRIPTION:
The Maternal Attachment Inventory (MAI) measure maternal love attachment (9). Muller tested the MAI questions in two phases; maternal adaptation and maternal attachmentEach item is evaluated by a 4-way to 26-point Likert-type scale ranging from "always" to "never". Always is calculated as (a) = 4 points, often (b) = 3 points, sometimes (c) = 2 points and never (d) = 1 point. The lowest score which could be obtained from the scale that measures maternal emotions and behaviors indicating love is 26, the high score is 104, and a high score indicates a high maternal attachment (12).

ELIGIBILITY:
Inclusion Criteria:

* natural pregnancy (without any Assisted reproductive technology (ART) method)
* aged 18 to 45 years
* no adverse obstetric history

Exclusion Criteria:

* psychiatric diagnosis
* history of psychiatric drug use
* postpartum blues
* known complications during pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Two hundred patients were divided into two groups. 100 women delivered vaginally and another 100 delivered with cesarean section. They were examined three month after delivery using Maternal Attachment Inventory (MAI) and a detailed history was taken.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Compare mother-infant bond (MIB) scores between the vaginal delivery and the C-section (C/S) groups. | 3 months
  They were examined three month after delivery using Maternal Attachment Inventory (MAI); Each item is evaluated by a 4-way to 26-point Likert-type scale ranging from "always" to "never". Always is calculated as (a) = 4 points, often (b) = 3 points, sometimes (c) = 2 points and never (d) = 1 point. The lowest score which could be obtained from the scale that measures maternal emotions and behaviors indicating love is 26, the high score is 104, and a high score indicates a high maternal attachment

SECONDARY OUTCOMES:
evaluate the correlations between the MIB scores and their sociodemographic data. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes